CLINICAL TRIAL: NCT00560066
Title: A Phase IV, Multi-Center, Active-Controlled, Observer-Blind Study to Evaluate the Safety of a Trivalent Subunit Influenza Vaccine Produced Either in Mammalian Cell Culture (Optaflu®) or in Embryonated Hen Eggs (Agrippal®) in Adults and Elderly With and Without Underlying Medical Conditions, and to Evaluate the Immunogenicity in a Subset of Subjects With Underlying Medical Conditions
Brief Title: Safety of a Influenza Vaccine Produced Either in Mammalian Cell Culture or in Embryonated Hen Eggs in Adults and Elderly With and Without Underlying Medical Conditions, and Immunogenicity in a Subset of Subjects With Underlying Medical Conditions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: V58P14; 2007-002872-32
Record Dates: First submitted 2007-11-16; First posted 2007-11-19 (Estimated); Results first posted 2013-04-18 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-01

CONDITIONS: Seasonal Influenza; Vaccine
Keywords: influenza; vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- cTIV (Experimental): Subjects received one vaccination of cell culture-derived influenza vaccine
  Interventions: Biological: Cell-derived influenza vaccine
- TIV (Active Comparator): Subjects received one vaccination of egg-derived influenza vaccine
  Interventions: Biological: Egg-derived influenza vaccine

INTERVENTIONS:
Biological: Cell-derived influenza vaccine — 1 dose of 0.5 mL in the deltoid region of the non-dominant arm
  Arms: cTIV
Biological: Egg-derived influenza vaccine — 1 dose of 0.5 mL in the deltoid region of the non-dominant arm
  Arms: TIV

SUMMARY:
Evaluation of the safety of Trivalent Subunit Influenza Vaccine Produced either in Mammalian Cell Culture or in embryonated Hen Eggs in subjects 18 years of age and above with and without underlying medical conditions and evaluation of the immunogenicity in a subset of subjects with underlying medical conditions, compared to an egg-based vaccine in a post marketing setting.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects 18 years of age and above, mentally competent, willing and able to give informed consent prior to study entry;
2. Able to comply with all study procedures and requirements.

Exclusion Criteria:

1. History of any anaphylaxis, serious vaccine reactions, or hypersensitivity to any vaccine component;
2. Fatal prognosis of an underlying medical condition (<12 months life expectancy);
3. History of Guillain-Barre syndrome;
4. Bleeding diathesis or receiving anticoagulants of the coumarin type;
5. Hospitalization or residence in a nursing care facility;
6. Planned to receive seasonal influenza vaccine outside of this study;
7. Receipt of another vaccine within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study;
8. Fever (defined as axillary temperature ≥38.0°C) or any acute illness within 3 days prior to study vaccination;
9. Receipt of another investigational agent within 30 days prior to enrollment in the study or before completion of the safety follow-up period in another study, whichever is longer, and unwilling to refuse participation in another clinical study through the end safety follow up period of the study;
10. Any condition, which, in the opinion of the investigator, might prevent the subject from participation or interfere with the evaluation of the study objectives;
11. Females who were pregnant or nursing (breastfeeding) mothers, or females of childbearing potential who were sexually active and had not used or did not plan to use acceptable birth control measures during the first 3 weeks after vaccination. Oral, injected or implanted hormonal contraceptive, diaphragm or condom with spermicidal agent or intrauterine device were considered acceptable forms of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1398 (Actual)
Dates: Start 2007-11; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (15):
- Germany (15):
  - Balve
  - Duisberg
  - Garmisch-Partenkirchen
  - Hanover
  - Herborn
  - Illingen
  - Kiel
  - Laufach
  - Marburg
  - Midlum
  - Olpe
  - Potsdam
  - Regensburg
  - Unterschleissheim
  - Wiesbaden

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 17 centres in Germany.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- Egg-derived Vaccine (TIV): Subjects received one vaccination of a egg-derived trivalent influenza virus vaccine.
- Cell Culture-derived Vaccine (cTIV): Subjects received one vaccination of a cell-derived trivalent influenza virus vaccine.
Period: Overall Study
Arm/Group | Egg-derived Vaccine (TIV) | Cell Culture-derived Vaccine (cTIV)
Started | 396 | 1002
Completed | 390 | 980
Not Completed | 6 | 22
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 4 | 10
Not completed — Protocol Violation | 0 | 1
Not completed — Administrative reason | 0 | 5
Not completed — Missing primary reason | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Egg-derived Vaccine (TIV) | Cell Culture-derived Vaccine (cTIV) | Total
Number analyzed (Participants) | 396 | 1002 | 1398
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (17.3) | 48.7 (16.3) | 48.3 (16.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206 | 533 | 739
  Male | 190 | 469 | 659

OUTCOME MEASURES:

1. Secondary Outcome: Number of Healthy Adults and Elderly Who Reported Solicited Local and Systemic Adverse Events (AEs) After One Vaccination of TIV or cTIV
Description: Analysis was performed on a subset of safety population which included the healthy adults (≥18 to ≤60 years) and elderly (≥61 years).
Time Frame: From Day 1 through Day 7 post-vaccination
Population: Analysis was done on a subset of safety population (i.e. all subjects in the exposed population who provide postvaccination safety data) which included the healthy adults and elderly.
Measure: Number; unit: Subjects
Groups:
- TIV (Adults): Subjects ≥18 to ≤60 years years-old received one vaccination of egg-derived influenza virus vaccine
- cTIV (Adults): Subjects ≥18 to ≤60 years-old received one vaccination of cell-derived influenza virus vaccine
- TIV (Elderly): Subjects ≥61 years-old received one vaccination of egg-derived influenza virus vaccine
- cTIV (Elderly): Subjects ≥61 years-old received one vaccination of cell-derived influenza virus vaccine
Arm/Group | TIV (Adults) | cTIV (Adults) | TIV (Elderly) | cTIV (Elderly)
Number analyzed (Participants) | 70 | 235 | 7 | 11
Subjects
  Pain (N=66,226,7,11) | 24 | 107 | 1 | 2
  Chills (N=66,226,7,11) | 1 | 10 | 0 | 0
  Malaise (N=66,226,7,11) | 7 | 25 | 0 | 0
  Myalgia (N=66,226,7,11) | 10 | 46 | 0 | 0
  Arthralgia (N=66,226,7,11) | 2 | 13 | 0 | 1
  Headache (N=66,226,7,11) | 14 | 47 | 0 | 2
  Sweating (N=66,226,7,11) | 1 | 13 | 2 | 0
  Fatigue (N=66,226,7,11) | 11 | 49 | 1 | 1
  Fever (≥38 °C) | 0 | 2 | 0 | 0

2. Secondary Outcome: Number of Adults and Elderly With Underlying Medical Conditions Who Reported Solicited Local and Systemic Adverse Events After One Vaccination of TIV or cTIV
Description: Analysis was performed on a subset of safety population which included the adults (≥18 to ≤60 years) and elderly (≥61 years) with underlying medical conditions.
Time Frame: From Day 1 through Day 7 post-vaccination
Population: Analysis was done on the subset of safety population which included the adults and elderly with underlying medical conditions.
Measure: Number; unit: Subjects
Groups:
- TIV (Adults): Subjects ≥18 to ≤60 years-old received one vaccination of egg-derived influenza virus vaccine
Arm/Group | TIV (Adults) | cTIV (Adults) | TIV (Elderly) | cTIV (Elderly)
Number analyzed (Participants) | 220 | 490 | 99 | 265
Subjects
  Pain (N=220,484,98,263) | 77 | 189 | 15 | 32
  Chills (N=220,484,98,263) | 5 | 15 | 3 | 9
  Malaise (N=220,484,98,263) | 27 | 51 | 5 | 13
  Myalgia (N=220,484,98,263) | 32 | 80 | 15 | 23
  Arthralgia (N=220,484,98,263) | 10 | 35 | 8 | 14
  Headache (N=220,484,98,263) | 40 | 94 | 15 | 40
  Sweating (N=220,484,98,263) | 12 | 33 | 6 | 10
  Fatigue (N=220,484,98,263) | 37 | 102 | 14 | 33
  Fever (≥38 °C) | 1 | 5 | 2 | 1

3. Secondary Outcome: Percentages Of Subjects With Underlying Medical Conditions Who Achieved Hemagglutination Inhibition (HI) Titer ≥40 After One Vaccination of TIV or cTIV
Description: Immunogenicity was measured as the percentage of adults (≥18 to ≤60 years) and elderly (≥61 years) achieving HI titers ≥40 at baseline (Day 1) and three weeks (Day 22) after one vaccination of TIV or cTIV for each of three vaccine strains, evaluated using hemagglutination inhibition (HI) egg-derived antigen assay. This criterion is met according to European (CHMP) guideline if the percentage of subjects achieving HI titers ≥40 is >70% (≥18 to ≤60 years), or >60% (≥61 years).
Time Frame: Before vaccination (Day 1) and three weeks after vaccination (Day 22)
Population: Analysis was performed on the immunogenicity subset of adults and elderly with underlying medical conditions (full analysis set [FAS]: all enrolled subjects who received a study vaccine and provided one evaluable serum sample before and after baseline)
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | TIV (Adults) | cTIV (Adults) | TIV (Elderly) | cTIV (Elderly)
Number analyzed (Participants) | 118 | 118 | 25 | 25
Percentages of Subjects
  A/H1N1 (Day 1) | 56 [46 to 65] | 53 [43 to 62] | 40 [21 to 61] | 56 [35 to 76]
  A/H1N1 (Day 22) | 98 [94 to 100] | 95 [89 to 98] | 96 [80 to 100] | 100 [86 to 100]
  A/H3N2 (Day 1) | 53 [44 to 63] | 46 [37 to 55] | 80 [59 to 93] | 64 [43 to 82]
  A/H3N2 (Day 22) | 97 [92 to 99] | 87 [80 to 93] | 100 [86 to 100] | 88 [69 to 97]
  B (Day 1) | 14 [8 to 21] | 16 [10 to 24] | 40 [21 to 61] | 28 [12 to 49]
  B (Day 22) | 77 [68 to 84] | 63 [53 to 71] | 68 [46 to 85] | 48 [28 to 69]

4. Secondary Outcome: Percentages Of Subjects Who Achieved Seroconversion Or Significant Increase In HI Titers After One Vaccination of TIV or cTIV
Description: Seroconversion or significant increase in HI titer as per CHMP criteria for each of the three strains is defined as the percentage of subjects with a prevaccination HI titer <10 to a postvaccination titer ≥40; or in subjects with prevaccination HI titer ≥10, a ≥4-fold increase in postvaccination HI antibody titer. According to the CHMP criteria, the percentage of subjects achieving seroconversion/significant increase should be >40% (≥18 to ≤60 years) or >30% (≥61 years).
Time Frame: Three weeks post-vaccination (Day 22)
Population: Analysis was performed on the immunogenicity subset of adults and elderly with underlying medical conditions.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | TIV (Adults) | cTIV (Adults) | TIV (Elderly) | cTIV (Elderly)
Number analyzed (Participants) | 118 | 118 | 25 | 25
Percentages of Subjects
  A/H1N1 | 64 [54 to 72] | 65 [56 to 74] | 72 [51 to 88] | 60 [39 to 79]
  A/H3N2 | 62 [52 to 71] | 56 [46 to 65] | 40 [21 to 61] | 40 [21 to 61]
  B | 55 [46 to 64] | 41 [32 to 50] | 24 [9 to 45] | 20 [7 to 41]

5. Secondary Outcome: Geometric Mean Titers of Subjects With Underlying Medical Conditions After One Vaccination of TIV or cTIV
Description: Immunogenicity was measured as HI geometric mean titers (GMTs) of subjects with underlying conditions, directed against each of three vaccine strains at baseline (Day 1) and three weeks after vaccination (Day 22) in adults (≥18 to ≤60 years) and elderly (≥61 years).
Time Frame: Before vaccination (Day 1) and three weeks after vaccination (Day 22)
Population: Analysis was performed on the immunogenicity subset of adults and elderly with underlying medical conditions.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | TIV (Adults) | cTIV (Adults) | TIV (Elderly) | cTIV (Elderly)
Number analyzed (Participants) | 118 | 118 | 25 | 25
Titers
  A/H1N1 (Day 1) | 37 [27 to 49] | 34 [25 to 46] | 19 [11 to 33] | 29 [17 to 51]
  A/H1N1 (Day 22) | 354 [282 to 443] | 308 [246 to 386] | 132 [87 to 199] | 158 [104 to 238]
  A/H3N2 (Day 1) | 31 [23 to 40] | 29 [22 to 38] | 56 [32 to 97] | 41 [23 to 71]
  A/H3N2 (Day 22) | 224 [179 to 281] | 156 [125 to 196] | 174 [112 to 271] | 145 [93 to 226]
  B (Day 1) | 9.35 [7.96 to 11] | 11 [9.24 to 13] | 20 [13 to 31] | 14 [8.86 to 21]
  B (Day 22) | 55 [46 to 66] | 39 [32 to 47] | 43 [26 to 72] | 26 [16 to 44]

6. Secondary Outcome: Geometric Mean Ratio of Subjects With Underlying Medical Conditions After One Vaccination of TIV or cTIV
Description: Immunogenicity was measured as the geometric mean ratio (GMR), calculated as the ratio of postvaccination to prevaccination HI GMTs for each of the three strains, three weeks after one vaccination (Day 22) of TIV or cTIV. CHMP criteria is considered fulfilled for each of the three strains if the geometric mean increase GMR (Day 22/Day 1) in HI antibody titer is >2.5 (≥18 to ≤60 years) or >2.0 (≥61 Years).
Time Frame: Three weeks post-vaccination (Day 22)
Population: Analysis was performed on the immunogenicity subset of adults and elderly with underlying medical conditions.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | TIV (Adults) | cTIV (Adults) | TIV (Elderly) | cTIV (Elderly)
Number analyzed (Participants) | 118 | 118 | 25 | 25
Ratio
  A/H1N1 | 9.65 [7.03 to 13] | 9 [6.55 to 12] | 6.96 [3.98 to 12] | 5.35 [3.06 to 9.37]
  A/H3N2 | 7.35 [5.62 to 9.61] | 5.32 [4.07 to 6.95] | 3.12 [1.76 to 5.51] | 3.58 [2.02 to 6.33]
  B | 5.88 [4.62 to 7.49] | 3.57 [2.8 to 4.54] | 2.17 [1.3 to 3.64] | 1.92 [1.15 to 3.21]

7. Primary Outcome: Number of Subjects Who Reported At Least One Reactogenicity Sign After One Vaccination of TIV or cTIV
Description: Safety was assessed as the number of all subjects who reported at least one sign of reactogenicity after one vaccination of egg-derived (TIV) or cell culture-derived (cTIV) influenza virus vaccine from Day 1 through Day 7 post-vaccination.
Time Frame: From Day 1 up to and including Day 7 post-vaccination
Population: Analysis was performed on the safety dataset, i.e. all subjects in the exposed set who provided post-baseline safety data.
Measure: Number; unit: Subjects
Arm/Group | Egg-derived Vaccine (TIV) | Cell Culture-derived Vaccine (cTIV)
Number analyzed (Participants) | 396 | 1001
Subjects
  Any reaction - Missing | 1 | 2
  Any reaction - None | 204 | 488
  Any reaction - Other than severe | 186 | 495
  Any reaction - Severe | 5 | 16
  Local reaction - Missing | 5 | 17
  Local reaction - None | 274 | 654
  Local reaction - Other than severe | 117 | 325
  Local reaction - Severe | 0 | 5
  Systemic reaction - Missing | 1 | 2
  Systemic reaction - None | 250 | 616
  Systemic reaction - Other than severe | 140 | 369
  Systemic reaction - Severe | 5 | 14

ADVERSE EVENTS:
Time Frame: Throughout the study period (day 1 to day 181).
Description: All enrolled subjects met entry criteria with one exception. One subject was enrolled and randomized to the CTIV group but did not receive the study vaccine due to a protocol deviation. This subject was excluded from both the safety and immunogenicity analyses.
Arm/Group | Egg-derived Vaccine (TIV) | Cell Culture-derived Vaccine (cTIV)
Serious Adverse Events (participants affected / at risk) | 10/396 | 20/1001
Other Adverse Events (participants affected / at risk) | 204/396 | 568/1001
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Egg-derived Vaccine (TIV) (N=396) | Cell Culture-derived Vaccine (cTIV) (N=1001)
Acute Chest Syndrome (Blood and lymphatic system disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 0
Aortic Valve Incompetence (Cardiac disorders) | 0 | 1
Aortic Valve Stenosis (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Sudden Hearing Loss (Ear and labyrinth disorders) | 0 | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Device Occlusion (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Device Related Infection (Infections and infestations) | 0 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Otitis Media (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 2
Urinary Tract Infection (Infections and infestations) | 1 | 1
Animal Bite (Injury, poisoning and procedural complications) | 0 | 1
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 1
Optic Neuritis (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient Ischaemic Attack (Nervous system disorders) | 1 | 1
Urethral Caruncle (Renal and urinary disorders) | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Deep Vein Thrombosis (Vascular disorders) | 1 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Egg-derived Vaccine (TIV) (N=396) | Cell Culture-derived Vaccine (cTIV) (N=1001)
Fatigue (General disorders) | 63 | 185
Injection site pain (General disorders) | 117 | 330
Malaise (General disorders) | 39 | 89
Bronchitis (Infections and infestations) | 14 | 59
Nasopharyngitis (Infections and infestations) | 10 | 90
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 76
Myalgia (Musculoskeletal and connective tissue disorders) | 57 | 150
Headache (Nervous system disorders) | 73 | 198
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 21 | 56

LIMITATIONS AND CAVEATS:
Because cTIV was not available, the second part of the study was not performed. In addition, as deviations from protocol procedures and GCP were identified at some sites, data collected for this study were not used to support licensure of cTIV.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No